CLINICAL TRIAL: NCT05511428
Title: Open Label Single Arm Study to Assess the Implementation of Home Based Daratumumab Administration in Patients Being Treated for Multiple Myeloma
Brief Title: Home Based Daratumumab Administration for Patients With Multiple Myeloma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22C.210; JT 19521 (Other: JeffTrial Number)
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab and hyaluronidase-fihj) (Experimental): Patients receive daratumumab and hyaluronidase-fihj SC over 3-5 minutes in the infusion center on day 1 of cycles 1, 2, 7, and 8 and at home on day 1 of cycles 3, 4, 5, and 6. Cycles repeat every 28 days for 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Daratumumab and Hyaluronidase-fihj; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Other: Interview

INTERVENTIONS:
Drug: Daratumumab and Hyaluronidase-fihj — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Interview — Ancillary studies

SUMMARY:
This clinical trial tests the treatment effect of home based daratumumab administration in treating patients with multiple myeloma. Darzalex Faspro is a combination of two drugs (daratumumab and hyaluronidase) used to treat adults with multiple myeloma. Daratumumab is in a class of medications called monoclonal antibodies. It works by helping the body to slow or stop the growth of cancer cells. Hyaluronidase-fihj is an endoglycosidase. It helps to keep daratumumab in the body longer so that the medication will have a greater effect. Standard medical care requires Darzalex-Faspro treatment be administered during visits to the cancer center. Receiving medication in the home setting, may decrease cost and burden of care in patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate treatment burden (using the Cancer Treatment Satisfaction Questionnaire [CTSQ]).

SECONDARY OBJECTIVES:

I. Determine adherence to home delivery of daratumumab and hyaluronidase-fihj (darzalex faspro).

II. Evaluate quality of life (using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ-30]) based on site of care (home versus [vs.] infusion center).

III. Evaluate financial burden (using the COST survey) based on site of care (home vs. infusion center).

IV. Evaluate Safety of home administration of darzalex-faspro. V. Evaluate barriers to home administration.

EXPLORATORY OBJECTIVES:

I. Evaluate patient perceptions of home administration of anti-neoplastic therapy.

II. Evaluate opportunity cost based on site of care (home vs. infusion center) (using the Oncology Opportunity Cost Assessment Tool [OOCAT] survey).

OUTLINE:

Patients receive daratumumab and hyaluronidase-fihj subcutaneously (SC) over 3-5 minutes in the infusion center on day 1 of cycles 1, 2, 7, and 8 and at home on day 1 of cycles 3, 4, 5, and 6. Cycles repeat every 28 days for 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged greater than 18 years of age
* Has a diagnosis of Multiple Myeloma
* Is on the monthly phase of daratumumab (either intravenous [IV] or subcutaneous [SubQ]) based regimen (every 4 weeks) (either monotherapy or in combination with oral agents)
* Is willing to receive daratumumab subcutaneous injections
* Lives within the range of Jefferson Home Infusion Services
* Patients are willing to allow home infusion company visit them and administer Darzalex-Faspro in the home
* Women of reproductive potential must use highly effective contraception
* Men of reproductive potential must use highly effective contraception
* Absolute neutrophil count (ANC) > 1,000
* Platelet count > 50,000
* Aspartate aminotransferase (AST) / alanine transaminase (ALT) < 2.5 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine clearance (CrCl) >= 20 mL/min for single agent subcutaneous (SC) daratumumab. For combination studies: with lenalidomide >= 30 mL/min
* English speaking

Exclusion Criteria:

* Receiving daratumumab for an indication other than multiple myeloma
* Receiving daratumumab in combination with other IV or subcutaneous therapy
* Pregnancy or lactation
* Known allergic reactions to components of the study product(s)
* Uncontrolled human immunodeficiency virus (HIV)
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]) who are not on hepatitis B prophylaxis. Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive and not on Hep B prophylaxis will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV deoxyribonucleic acid (DNA) by PCR
* Patients with reactivation of hepatitis B will be excluded
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as a viremia at least 12 weeks after completion of antiviral therapy)
* Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal
* Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate
* Clinically significant cardiac disease, including:

  * Myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
  * Uncontrolled cardiac arrhythmia
  * Screening 12-lead electrocardiogram (ECG) showing a baseline QT interval as corrected by Fridericia's formula > 470 msec
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam R Binder, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Daratumumab and Hyaluronidase-fihj)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 1
Description: Treatment satisfaction was assessed using the Satisfaction with Therapy (SWT) subscale of the Cancer Treatment Satisfaction Questionnaire (CTSQ). The Cancer Therapy Satisfaction Questionnaire (CTSQ) measures a patient's satisfaction with cancer treatment across several domains. The SWT score ranges from 0 to 100, where a higher score represents a better outcome, indicating greater satisfaction or fewer issues. Results are represented as the mean SWT score and the standard deviation (SD) at each specified cycle.
Time Frame: At Visit 1,Baseline
Population: Although 20 participants were enrolled in the study, not all participants completed the CTSQ at each time point. As a result, only the 19 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-100) | 87.2 (10.5)

2. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 2
Description: as for outcome 1
Time Frame: At Visit 2, Day29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-100) | 87.4 (7.9)

3. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 3
Description: as for outcome 1
Time Frame: At Visit 3, Day 57
Population: Although 20 participants were enrolled in the study, not all participants completed the CTSQ at each time point. As a result, only the 18 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 18
scores on a scale (0-100) | 89.3 (10.2)

4. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 4
Description: as for outcome 1
Time Frame: At Visit 4, Day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-100) | 86.1 (10.3)

5. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 5
Description: as for outcome 1
Time Frame: At Visit 5, Day 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-100) | 88.2 (9.5)

6. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 6
Description: as for outcome 1
Time Frame: At Visit 6, Day 141
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 18
scores on a scale (0-100) | 85.7 (14.1)

7. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 7
Description: as for outcome 1
Time Frame: At Visit 7, Day 169
Population: Although 20 participants were enrolled in the study, not all participants completed the CTSQ at each time point. As a result, only the 16 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 16
scores on a scale (0-100) | 89.7 (11.8)

8. Primary Outcome: Treatment Satisfaction Will be Measured Using the SWT Score From the Cancer Treatment Satisfaction Questionnaire (CTSQ) - Cycle 8
Description: as for outcome 1
Time Frame: At Visit 8, Day 197
Population: Although 20 participants were enrolled in the study, not all participants completed the CTSQ at each time point. As a result, only the 17 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 17
scores on a scale (0-100) | 90.1 (12.7)

9. Secondary Outcome: Number of Participants With Medication Adherence in Home Setting During Cycle 3
Description: Adherence is defined as completing administration of medication in the home setting during cycles 3-6. Adherence will be measured for each dose given and failure would occur if the participant needs to go to the infusion center for administration for whatever reason. Based on previous studies of home based administration adherence rates over 75% would be needed to meet criteria for feasibility. The adherence at the home setting cycles will be analyzed in repeated measures logistic regression model with a random effect of patient and the fixed effect of the delivery mode (home vs. infusion center).
Time Frame: At Visit 3,Day 57
Population: Participants who received at least one dose in the home setting during cycle 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 19

10. Secondary Outcome: Number of Participants With Medication Adherence in Home Setting During Cycle 4
Description: as for outcome 9
Time Frame: At Visit 4,Day 85
Population: Participants who received at least one dose in the home setting during cycle 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 19

11. Secondary Outcome: Number of Participants With Medication Adherence in Home Setting During Cycle 5
Description: as for outcome 9
Time Frame: At Visit 5,Day 113
Population: Participants who received at least one dose in the home setting during cycle 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 19

12. Secondary Outcome: Number of Participants With Medication Adherence in Home Setting During Cycle 6
Description: as for outcome 9
Time Frame: At Visit 6,Day 141
Population: Participants who received at least one dose in the home setting during cycle 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 19

13. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 1
Description: Global Health Status was assessed using the Global Health Status/QoL subscale of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-30). Scores range from 0-100, with higher scores indicating better global health status and quality of life. Results represent the mean Global Health Status/QoL score and standard deviation (SD) for each arm at the specified cycle.
Time Frame: At Visit 1, Baseline
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 20
scores on a scale (0-100) | 64.2 (21.3)

14. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 2
Description: as for outcome 13
Time Frame: At Visit 2, Day 29
Population: Although 20 participants were enrolled in the study, not all participants completed the EORTC QLQ-30 at each time point. As a result, only the 19 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-100) | 69.3 (17.4)

15. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 3
Description: as for outcome 13
Time Frame: At Visit 3, Day 57
Population: Although 20 participants were enrolled in the study, not all participants completed the EORTC QLQ-30 at each time point. As a result, only the 18 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 18
scores on a scale (0-100) | 64.4 (15.9)

16. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 4
Description: as for outcome 13
Time Frame: At Visit 4, Day 85
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-100) | 65.8 (19.6)

17. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 5
Description: as for outcome 13
Time Frame: At Visit 5, Day 113
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-100) | 57.5 (18.4)

18. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 6
Description: as for outcome 13
Time Frame: At Visit 6, Day 141
Population: Although 20 participants were enrolled in the study, not all participants completed the EORTC QLQ-30 at each time point. As a result, only the 17 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 17
scores on a scale (0-100) | 69.1 (20.8)

19. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 7
Description: as for outcome 13
Time Frame: At Visit 7, Day 169
Population: Although 20 participants were enrolled in the study, not all participants completed the EORTC QLQ-30 at each time point. As a result, only the 16 participants who provided complete and analyzable responses were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 16
scores on a scale (0-100) | 69.3 (18.4)

20. Secondary Outcome: Global Health Status/Quality of Life Score (EORTC QLQ-30) At Cycle 8
Description: as for outcome 13
Time Frame: At Visit 8, Day 197
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: scores on a scale (0-100)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 17
scores on a scale (0-100) | 62.3 (18.9)

21. Secondary Outcome: Financial Toxicity
Description: Financial toxicity will be measured using the COST survey. FACIT-COST (v2) score (range: 0-44). A lower score indicates higher financial toxicity, while a higher score implies better financial well-being.
Time Frame: At Visit 1, Baseline
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-44) | 27.0 (7.8)

22. Secondary Outcome: Financial Toxicity
Description: as for outcome 21
Time Frame: At Visit 2, Day 29
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-44) | 28.5 (9.9)

23. Secondary Outcome: Financial Toxicity
Description: as for outcome 21
Time Frame: At Visit 3, Day 57
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 18
scores on a scale (0-44) | 24.8 (9.7)

24. Secondary Outcome: Financial Toxicity
Description: as for outcome 21
Time Frame: At Visit 4, Day 85
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-44) | 28 (9.2)

25. Secondary Outcome: Financial Toxicity
Description: as for outcome 21
Time Frame: At Visit 5, Day 113
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
scores on a scale (0-44) | 26.8 (10.4)

26. Secondary Outcome: Financial Toxicity
Description: as for outcome 21
Time Frame: At Visit 6, Day 141
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 17
scores on a scale (0-44) | 26.6 (10.4)

27. Secondary Outcome: Financial Toxicity
Description: as for outcome 21
Time Frame: At Visit 7, Day 169
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 16
scores on a scale (0-44) | 24.7 (9.6)

28. Secondary Outcome: Financial Toxicity
Description: as for outcome 21
Time Frame: At Visit 8, Day 197
Measure: Mean (Standard Deviation); unit: scores on a scale (0-44)
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 17
scores on a scale (0-44) | 27.7 (9.0)

29. Secondary Outcome: Number of Adverse Events During Home Administration
Description: Safety will be evaluated through collection of adverse events. Total number of adverse events occurring more than 1% of the time that occured during cycle 3-6, when Darzalex-Faspro was administered at home.
Time Frame: Cycle 3 through Cycle 6, days 57-169
Population: All participants who received Darzalex-Faspro during specified cycles.
Measure: Number; unit: adverse events
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
adverse events | 69

30. Secondary Outcome: Number of Adverse Events During Infusion Center Administration
Description: Safety will be evaluated through collection of adverse events. Total number of adverse events that occurred more than 1% of the time during cycles 1, 2, 7, and 8 when Darzalex-Faspro was administered at the infusion center.
Time Frame: Cycle 1, Cycle 2, Cycle 7, and Cycle 8, days 1-57 and 169-197
Population: All participants who received Darzalex-Faspro during specified cycles.
Measure: Number; unit: adverse events
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
adverse events | 82

31. Secondary Outcome: Number of Patients Reporting Barriers to Home Administration At Cycle 3
Description: Barriers to receiving home administration were assessed using binary (yes/no) questionnaire administered at Cycle 3. Participants were asked whether they experienced any barriers to home infusion, including delays in treatment related to delivery of medication, arrival time of the infusion nurse, issues related to storage of medication, issues related to administration of the medication. The outcome reflects the total number of participants who responded, "yes" to any barriers to home based therapy, based on binary (yes/no) questionnaire.
Time Frame: At Visit 3, Day 57
Population: All participants who received Darzalex-Faspro in the home setting during cycles 3-6.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 0

32. Secondary Outcome: Number of Patients Reporting Barriers to Home Administration At Cycle 4
Description: Barriers to receiving home administration were assessed using binary (yes/no) questionnaire administered at Cycle 4. Participants were asked whether they experienced any barriers to home infusion, including delays in treatment related to delivery of medication, arrival time of the infusion nurse, issues related to storage of medication, issues related to administration of the medication. The outcome reflects the total number of participants who responded, "yes" to any barriers to home based therapy, based on binary (yes/no) questionnaire.
Time Frame: At Visit 4, Day 85
Population: All participants who received Darzalex-Faspro in the home setting during cycles 3-6.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 0

33. Secondary Outcome: Number of Patients Reporting Barriers to Home Administration At Cycle 5
Description: Barriers to receiving home administration were assessed using binary (yes/no) questionnaire administered at Cycle 5. Participants were asked whether they experienced any barriers to home infusion, including delays in treatment related to delivery of medication, arrival time of the infusion nurse, issues related to storage of medication, issues related to administration of the medication. The outcome reflects the total number of participants who responded, "yes" to any barriers to home based therapy, based on binary (yes/no) questionnaire.
Time Frame: At Visit 5, Day 113
Population: All participants who received Darzalex-Faspro in the home setting during cycles 3-6.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 0

34. Secondary Outcome: Number of Patients Reporting Barriers to Home Administration At Cycle 6
Description: Barriers to receiving home administration were assessed using binary (yes/no) questionnaire administered at Cycle 6. Participants were asked whether they experienced any barriers to home infusion, including delays in treatment related to delivery of medication, arrival time of the infusion nurse, issues related to storage of medication, issues related to administration of the medication. The outcome reflects the total number of participants who responded, "yes" to any barriers to home based therapy, based on binary (yes/no) questionnaire.
Time Frame: At Visit 6, Day 141
Population: All participants who received Darzalex-Faspro in the home setting during cycles 3-6. No barriers were identified.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants | 0

35. Other Pre Specified Outcome: Patient Perceptions of Home Based Anti-neoplastic Therapy
Description: Patient perceptions of home based anti-neoplastic therapy will be measured through semi-structured interviews.
Time Frame: Cycle 3 through Cycle 6, days 57-169
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 19
Participants
  Positive : Familiarity | 2
  Positive : Overall Comfort | 3
  Positive : Ability to Rest After Treatment | 3
  Positive : More Time in the Day for Work/Other Activities | 3
  Positive : Eliminated Travel Inconveniences | 3
  Positive : Acceptability of Home Blood Draws | 2
  Positive : Satisfaction with Home Infusion Staff | 2
  Negative : Wait Times | 6

36. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 1, Baseline
Population: Surveys were collected using the Oncology Opportunity Cost Assessment Tool (OOCAT) during the home administration period. However, the data could not be analyzed due to incorrectly completed responses. As a result, no summary statistics or conclusions could be drawn from the opportunity cost data.
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

37. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 2, Day 29
Population: as for outcome 36
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

38. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 3, Day 57
Population: as for outcome 36
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

39. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 4, Day 85
Population: as for outcome 36
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

40. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 5, Day 113
Population: as for outcome 36
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

41. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 6, Day 141
Population: as for outcome 36
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

42. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 7, Day 169
Population: as for outcome 36
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

43. Other Pre Specified Outcome: Opportunity Cost
Description: Opportunity cost will be measured through the Oncology Opportunity Cost Assessment Tool (OOCAT) survey.
Time Frame: At Visit 8, Day 197
Population: as for outcome 36
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The PI will follow adverse events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation, an average of 8 months. At each study visit, the investigator (or designee) will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization.
Arm/Group | Treatment (daratumumab and hyaluronidase-fihj)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (daratumumab and hyaluronidase-fihj) (N=20)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
stomach pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (daratumumab and hyaluronidase-fihj) (N=20)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Dental carriers (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Edema- limbs (General disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Fatigue (General disorders) | 8 (9)
Fever (General disorders) | 1 (1)
Flue like symptoms (General disorders) | 5 (5)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders- other (Gastrointestinal disorders) | 1 (1) — blood in vomit
Headache (Nervous system disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
infections and infestations- other (Infections and infestations) | 1 (1) — vertebral osteomyelitis discitis with epidural abscess
infusion related reaction (zometa) (Infections and infestations) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Metabolism and nutrition disorders- other (Metabolism and nutrition disorders) | 1 (1) — Vitamin B-12 deficiency
mucositis- oral (Gastrointestinal disorders) | 1 (1)
muscle cramp (Musculoskeletal and connective tissue disorders) | 4 (4)
muscle weakness- lower limbs (Musculoskeletal and connective tissue disorders) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified- other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Benign prostatic hyperplasia
Neoplasms benign, malignant and unspecified- other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — bladder mass
non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (pain in lower jaw) (Gastrointestinal disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9)
Paresthesia (Nervous system disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Teeth grinding
Peripheral sensory neuropathy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 2 (2)
rectal ulcer (Gastrointestinal disorders) | 1 (1)
sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous disorders- other (Skin and subcutaneous tissue disorders) | 1 (1) — rash over leg, seems like bruising from seam of pants
Skin and subcutaneous disorders- other (Skin and subcutaneous tissue disorders) | 1 (1) — rash, drug eruption
Skin and subcutaneous disorders- other (Skin and subcutaneous tissue disorders) | 1 (1) — bilateral atopic dermatitis of the ear
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
skin infection (Infections and infestations) | 1 (1)
stomach pain (Gastrointestinal disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 5 (5)
urinary frequency (Renal and urinary disorders) | 2 (2)
urinary tract infection (Infections and infestations) | 1 (1)
vascular disorders- other (Vascular disorders) | 1 (1) — abnormal vision, floaters in the left eye, thinning of blood vessels
viremia (Infections and infestations) | 1 (1)
vision decreased (Eye disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (3)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT05511428/Prot_SAP_000.pdf